CLINICAL TRIAL: NCT05934305
Title: Mitigating the Impact of Stigma and Shame as a Barrier to Viral Suppression Among People Living With HIV and Substance Use Disorders
Brief Title: Mitigating the Impact of Stigma and Shame Among People Living With HIV and Substance Use Disorders
Acronym: MATTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-44770; R01DA057298 (NIH)
Record Dates: First submitted 2023-06-20; First posted 2023-07-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hiv; Substance Use Disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matter Intervention (Experimental): This 5-session text-enhanced intervention is designed to mitigate the negative behavioral consequences of internalized stigma and shame among individuals with SUDs that perpetuate sub-optimal engagement in HIV self-care and consequently inconsistent viral suppression. The intervention involves five virtually delivered one-on-one therapy sessions focused on behavioral goal setting skill development and related self-efficacy, increasing meta-cognitive awareness (i.e., non-judgmental awareness of emotions and cognitions), and teaching and reinforcing compassionate self-restructuring (i.e., self-compassion). Participants also receive daily text messages querying emotions during the one-on-one portion of the intervention. For eight weeks after the one-on-one portion, participants receive their compassionate self-statements via text in response to their indicated emotions. Participants will also receive phone-based resource navigation, as needed.
  Interventions: Behavioral: Matter Intervention
- Control Condition (Active Comparator): The control condition will involve five sessions of prerecorded asynchronous content related to local resources (e.g., information related to substance use treatment and other ancillary services).
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Matter Intervention — This 5-session text-enhanced intervention is designed to mitigate the negative behavioral consequences of internalized stigma and shame among individuals with SUDs that perpetuate sub-optimal engagement in HIV self-care and consequently inconsistent viral suppression. The intervention involves five virtually delivered one-on-one therapy sessions focused on behavioral goal setting skill development and related self-efficacy, increasing meta-cognitive awareness (i.e., non-judgmental awareness of emotions and cognitions), and teaching and reinforcing compassionate self-restructuring (i.e., self-compassion). Participants also receive daily text messages querying emotions during the one-on-one portion of the intervention. For eight weeks after the one-on-one portion, participants receive their compassionate self-statements via text in response to their indicated emotions. Participants will also receive phone-based resource navigation, as needed.
  Arms: Matter Intervention
Behavioral: Control Condition — The control condition will involve five sessions of prerecorded asynchronous content related to local resources (e.g., information related to substance use treatment and other ancillary services).
  Arms: Control Condition

SUMMARY:
People living with HIV and substance use disorders (SUDs) are less likely to be virally suppressed, which can lead to HIV transmission and negative health outcomes. This hybrid type 1 study will assess the efficacy, mechanisms, as well as facilitators and barriers to implementing the MATTER intervention, a virtually delivered 5-session text-enhanced psychobehavioral intervention designed to facilitate viral suppression by addressing internalized stigma and shame as barriers to engagement in HIV care among individuals living with HIV and SUDs in two locations with different levels of HIV resources (i.e., the Boston, Massachusetts and Miami, Florida metro areas). MATTER aims to mitigate the negative behavioral consequences of internalized stigma and shame on viral suppression by a) developing behavioral self-care goal setting skills and related self-efficacy, b) increasing metacognitive awareness (i.e., non-judgmental awareness of emotions and cognitions), and c) teaching and reinforcing compassionate self-restructuring (i.e., self- compassion), in addition to providing access to phone-based resource navigation. Scalable interventions such as MATTER are essential to our efforts to end the HIV epidemic in high priority regions.

DETAILED DESCRIPTION:
Among individuals living with HIV, substance use disorders (SUDs) are associated with inadequate engagement in HIV care, often leading to episodic unsuppressed viral load (VL) or viral rebound, thus driving the epidemic through elevated HIV transmission risk. Behavioral science identifies that internalized stigmas perpetuated by negative experiences related to drug use and unmet needs influences sub-optimal engagement in HIV care, resultant unsuppressed VL, and transmission among people with SUDs. Stigma and related emotions (e.g., shame) compromise health outcomes both directly (e.g., via sub-optimal adherence and appointment attendance) and indirectly (e.g., as obstacles to needed service engagement). Interventions are needed to address stigma and shame as obstacles to viral suppression among individuals living with HIV and SUDs. To meet this need, we developed, refined, and conducted a pilot RCT (K23DA043418) to assess the feasibility and acceptability of the MATTER intervention, an evidence- and community- informed psychobehavioral intervention to facilitate viral suppression by reducing the impact of internalized stigma and shame on engagement in HIV care among individuals with SUDs. The MATTER intervention aims to mitigate the negative behavioral consequences of internalized stigma and shame on viral suppression by a) behavioral self-care goal setting skills and related self-efficacy, b) increasing metacognitive awareness (i.e., non-judgmental awareness of cognitions and emotions), and c) compassionate self-restructuring (i.e., self- compassion). It involves 5- one-on-one virtual therapy sessions and bidirectional personalized text messaging to extend the impact of the intervention while using less interventionist time and phone-based resource navigation. The proposed hybrid type 1 efficacy-implementation study will use the RE-AIM framework to assess: 1) the efficacy of the MATTER intervention on viral suppression at the final 12-month follow up visit compared to a time-matched control arm using a fully powered randomized controlled trial (RCT; N=256), 2) the proposed mechanisms of the MATTER intervention to inform future interventions to mitigate the impact of stigma, and 3) facilitators and obstacles to the reach, adoption, implementation, and maintenance of the MATTER intervention to be conducted in two priority locations with key differences: the Boston, Massachusetts and Miami, Florida metro areas. Should the intervention be efficacious, and the innovative internalized stigma mitigation approach be confirmed, we will be well-positioned to leverage the identified facilitators and obstacles to implementing this intervention among people living with HIV and SUDs in a subsequent hybrid type 2 trial to assess the scalability, including a full cost-effectiveness assessment.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Meet criteria for an illicit (not solely including tobacco, cannabis, or alcohol) SUD
* Endorse internalized stigma related to HIV, substance use, sexual orientation, or gender-identity
* Unsuppressed HIV VL (>20 copies/mL).
* Provide informed consent in English
* Verbally communicate in English and read in English or Spanish
* Be ≥18 years old
* Provide evidence or documentation of HIV+ status
* Release HIV-related health records
* Have access to a cell phone with text capacity (study will supplement phones and plans as needed consistent with our pilot work).

Exclusion Criteria:

* Cisgender women
* Cisgender heterosexual men

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Viral Suppression at 12 month follow-up | 12 month follow up
  Compare the proportion of participants randomized to the intervention to the proportion of those randomized to the time-matched control condition who are virally suppressed at the 12 months follow up visit.

SECONDARY OUTCOMES:
Viral Suppression at 6 month follow-up | 6 month follow up
  Compare the proportion of participants randomized to the intervention to those randomized to the control condition who are virally suppression at the 6 months follow up visit.
Viral Suppression at 6 and 12 months | 6 and 12 months
  Compare the proportion of participants randomized to the intervention to those randomized to the control condition who are virally suppressed at both 6- and 12-month visits.
Internalized HIV Stigma Scale at 6 and 12 | 6 and 12 months
  Compare changes in self-reported mean scores between baseline and 6 and 12 month follow up visits. Response options to each question range from 0 = none of the time to 4 = all of the time, resulting in a mean response of between 0-4. Higher scores indicate greater internalized stigma.
Substance Use Severity based on clinical diagnostic interview | 12 months
  Categorically assess the severity of substance use disorder severity (no substance use disorder, mild, moderate, or severe) for each participant at baseline and the final 12-month followup. Investigators will then compare the proportion of participants with severe substance use disorder at final follow up compared to baseline as well as the proportion who reduced their severity between baseline and the final follow up in clinically among participants randomized to the intervention versus the control condition.
Visual Analogue Scale for Antiretroviral Adherence | 12 months
  Participants will be asked to report what percentage of their antiretroviral medication they have taken in the past 4 weeks on a scale of 0-100%.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Batchelder, PhD, MPH, Principal Investigator — CABU School of Medicine, Psychiatry
Locations (2):
- United States (2):
  - Florida International University, Miami, Florida
  - Fenway Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No